CLINICAL TRIAL: NCT02704962
Title: A Randomized, Double-blind, Comparison of the Efficacy and Safety of Olanzapine Versus Low-dose Olanzapine Plus Low-dose Trifluoperazine in the Treatment of Schizophrenia
Brief Title: Olanzapine vs. Low-dose Olanzapine Plus Trifluoperazine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Principal Investigator, Ching-Hua Lin, MD, PhD, Chief of Adult Psychiatry, Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSPH-2011-22
Record Dates: First submitted 2016-02-27; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; olanzapine; trifluoperazine; antipsychotic polypharmacy
MeSH Terms: conditions — Schizophrenia | interventions — Polypharmacy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trifluoperazine plus olanzapine (Experimental): trifluoperazine 5mg/day + olanzapine 5mg/day
  Interventions: Drug: full-dose olanzapine
- full-dose olanzapine (Active Comparator): olanzapine 10mg/day
  Interventions: Drug: full-dose olanzapine

INTERVENTIONS:
Drug: full-dose olanzapine — trifluoperazine 5mg/d
  Other Names: polypharmacy

SUMMARY:
The investigators hypothesis is that an antipsychotic drug combination of low-dose olanzapine plus low-dose trifluoperazine is similar to regular-dose olanzapine monotherapy in efficacy and safety for treatment of schizophrenia.The goal of this study is to compare the efficacy and safety of the olanzapine (10 mg/d) and olanzapine (5 mg/d) plus trifluoperazine (5 mg/d) in the treatment of acute psychotic exacerbations of schizophrenia.

DETAILED DESCRIPTION:
Antipsychotic monotherapy is recognized as the treatment of choice for patients with schizophrenia. Surveys have shown that antipsychotic polypharmacy are frequently prescribed, yet few randomized, double-blind clinical trials have examined this practice. Olanzapine, an atypical antipsychotic agent, has low incidence of extrapyramidal symptom but with high cost compared to trifluoperazine. It has been reported that mean doses of typical antipsychotics less than 600 mg per day of chlorpromazine or its equivalent has no higher risk of extrapyramidal symptom than atypical antipsychotics. The objective of the study is to compare the efficacy and safety of the olanzapine (10 mg per day) and olanzapine (5 mg per day) plus trifluoperazine (5 mg per day) in the treatment of acute psychotic exacerbations of schizophrenia. In this 6-week, double-blind, fixed-dose study, patients with schizophrenia are randomly assigned to olanzapine (10 mg per day)) or olanzapine (5 mg per day) plus trifluoperazine (5 mg per day). The hypothesis is that the two treatment groups have the similar efficacy and safety, but different cost. The primary efficacy measure is change from baseline in Positive and Negative Syndrome Scale (PANSS) total scores; secondary outcomes include Clinical Global Impression-Severity (CGI-S), the Calgary Depression Scale for Schizophrenia (CDSS), Global Assessment of Functioning Scale (GAF), Short Form-36 (SF-36), Mini Mental State Examination (MMSE). Safety assessments include the change from baseline on Simpson-Angus Rating Scale (SAS), Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS), and UKU Side-effects Rating Scale, and the change from baseline in prolactin levels, body weight, vital sign, blood pressure, Bazett's correction of QT interval (QTc interval), fasting glucose level, and lipid panel (cholesterol, high density lipid protein, low density lipid protein, and triglyceride).

ELIGIBILITY:
Inclusion Criteria:

* were physically healthy and had all laboratory parameters within normal limits
* were aged 18 to 55 years
* satisfied the DSM-IV criteria for schizophrenia
* had baseline Clinical Global Impression-Severity of Illness (CGI-S) scale score of 4 or greater
* had no DSM-IV diagnosis of substance abuse or dependence (including alcohol)
* had not received depot antipsychotic drugs for the preceding 3 months
* gave written informed consent to participate in the study after a full explanation of the study's aims and procedures.

Exclusion Criteria:

* those with a history of serious adverse reaction to olanzapine or trifluoperazine or a history of tardive dyskinesia or neuroleptic malignant syndrome
* female subjects who were pregnant or at risk for pregnancy or lactation
* those that had a diagnosis of treatment-resistant schizophrenia or having previously received clozapine or electroconvulsive therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2012-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The changes in the Positive and Negative Syndrome Scale (PANSS) scores from baseline to the end of the study. | The PANSS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).

SECONDARY OUTCOMES:
The changes in the Clinical Global Impression-Severity (CGI-S) scores from baseline to the end of the study. | The CGI-S was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Calgary Depression Scale for Schizophrenia (CDSS) scores from baseline to the end of the study. | The CDSS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Global Assessment of Functioning (GAF) scores from baseline to the end of the study. | The GAF was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Short-Form 36 (SF-36) scores from baseline to week 6. | The SF-36 was rated at baseline and again at week 6.
The changes in the Mini Mental State Examination (MMSE) scores from baseline to week 6. | The MMSE was rated at baseline and again at week 6.
The changes in the Simpson-Angus Rating Scale (SAS) scores from baseline to the end of the study. | The SAS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Abnormal Involuntary Movement Scale (AIMS) scores from baseline to the end of the study. | The AIMS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Barnes Akathisia Scale (BAS) scores from baseline to the end of the study. | The BAS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the UKU Side-effects Rating Scale (UKU) scores from baseline to the end of the study. | The UKU was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the Bazett's correction of QT interval (QTc interval) from baseline to week 6. | The QTc interval was assayed at baseline and again at week 6.
The changes in the body weight from baseline to the end of the study. | The body weight was assayed at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
The changes in the fasting glucose level from baseline to week 6. | The fasting glucose level was assayed at baseline and again at week 6.
The changes in the prolactin level from baseline to week 6. | The prolactin level was assayed at baseline and again at week 6.
The changes in the cholesterol level from baseline to week 6. | The cholesterol level was assayed at baseline and again at week 6.
The changes in the high density lipoprotein (HDL) level from baseline to week 6. | The HDL level was assayed at baseline and again at week 6.
The changes in the low density lipoprotein (LDL) level from baseline to week 6. | The LDL level was assayed at baseline and again at week 6.
The changes in the triglyceride level from baseline to week 6. | The triglyceride level was assayed at baseline and again at week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hua Lin, MD, PhD, Principal Investigator — Kaohsiung Municipal Kai-Syuan Psychiatric Hospital, Kaohsiung City, Taiwan; Cheng-Chung Cheng, MD, PhD, Study Chair — Kaohsiung Municipal Kai-Syuan Psychiatric Hospital, Kaohsiung City, Taiwan
Locations (1):
- Kai-Suan Psychiatric Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lin CH, Wang FC, Lin SC, Huang YH, Chen CC, Lane HY. Antipsychotic combination using low-dose antipsychotics is as efficacious and safe as, but cheaper, than optimal-dose monotherapy in the treatment of schizophrenia: a randomized, double-blind study. Int Clin Psychopharmacol. 2013 Sep;28(5):267-74. doi: 10.1097/YIC.0b013e3283633a83. PMID 23778382
- [Result] Leucht S, Corves C, Arbter D, Engel RR, Li C, Davis JM. Second-generation versus first-generation antipsychotic drugs for schizophrenia: a meta-analysis. Lancet. 2009 Jan 3;373(9657):31-41. doi: 10.1016/S0140-6736(08)61764-X. Epub 2008 Dec 6. PMID 19058842
- [Result] Lin CH, Kuo CC, Chou LS, Chen YH, Chen CC, Huang KH, Lane HY. A randomized, double-blind comparison of risperidone versus low-dose risperidone plus low-dose haloperidol in treating schizophrenia. J Clin Psychopharmacol. 2010 Oct;30(5):518-25. doi: 10.1097/JCP.0b013e3181f28dff. PMID 20814315